CLINICAL TRIAL: NCT04777799
Title: Effectiveness and Acceptability of a Digital Solution to Train Specific EEG Frequencies With Neurofeedback for Improving Sleep
Acronym: CONNECTOSOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of the sponsor
Sponsor: AdministrateurDRC (Other)
Collaborators: Urgotech (Industry); University Hospital, Grenoble (Other)
Responsible Party: Sponsor-Investigator, AdministrateurDRC, Pr, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC19.202; 2020-A02600-39 (Other: ID/RCB)
Record Dates: First submitted 2021-02-02; First posted 2021-03-02 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Insomnia; Sleep Disorder
Keywords: Insomnia; Neurofeedback
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, open-labelled, multicenter, French study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- URGOnight (Experimental): Use of the URGOnight neurofeedback training headband and its associated application
  Interventions: Device: URGOnight

INTERVENTIONS:
Device: URGOnight — URGOnight is a daytime brain training solution (CE marked) aim at improve the quality of sleep. The device consists of an electroencephalographic (EEG) measuring strip connected to a mobile application. The latter is available free of charge on Android and iOS in various mobile application stores (Google Play Store and App Store).
  URGOnight is a wireless device, it connects via Bluetooth® Low Energy (BLE) to the URGOnight mobile application running on a smartphone. The EEG data is broadcast via a BLE protocol, and the standard Bluetooth® operating distance has a range of 10 meters.
  To use the URGOnight solution, the user must authorize the application to access his phone's memory to store his usage data and must also authorize the geolocation of his phone to enable BLE connection. This data is not recorded but is necessary for the proper functioning of the solution.

SUMMARY:
The management of insomnia includes, as a first step, a healthy lifestyle, including physical activity at appropriate times, nutritional monitoring, reduced consumption of stimulants, bedtime and wake-up times that do not vary between weekdays and weekends, banning screens at least two hours before bedtime, etc. If all these conditions are met and insomnia persists, additionnal therapies may be offered. URGOTECH has developed a connected headband allowing to practice neurofeedback in complete autonomy in subjects reporting dissatisfaction with the quality of their sleep.

DETAILED DESCRIPTION:
Among the parameters of brain activity used in neurofeedback, the most frequently used EEG activity is training to strengthen sensorimotor rhythms (SMR). This training could make it possible to reduce cortical hyperstimulation associated with certain sleep disorders. Our hypothesis is that the application of such a neurofeedback technique in an ecological situation at home will improve the subjective quality of their sleep.

The subject must perform, at home, at least 3 sessions per week with the URGOnight solution for about 4 months. Since regularity is important in order to observe effects, subjects are followed up by smartphone application at least 3 times over the training period.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia according to DSM V criteria (sleep latency greater than or equal to 30 minutes, night-time waking time greater than 30 minutes and early awakening for at least 1 month)
* ISI score greater than or equal to 15
* Head circumference: 52-62 cm
* Subjects not suffering from a characterized depressive episode and/or severe anxiety (Hospital Anxiety and Depression Scale with Depression score<11 and Anxiety score<11)
* Having a smartphone (Android 5 or iOS 11), an internet connection and able to use it
* Able to give free, informed and written consent
* Affiliated or beneficiary of a social security

Exclusion Criteria:

* Organic Sleep Disorders: Sleep Apnea Syndrome, Restless Legs, Narcolepsy, Hypersomnia, Kleine-Levin, Sleep Related Eating Syndrome and Nocturnal Bulimia
* Acute or chronic pathologies incompatible with the study follow-up according to the investigator's assessment (severe psychiatric disorders by MMSE interview, acute pain and acute pain acutization)
* Antidepressants and/or hypnotics whose dosage was changed within 3 months prior to inclusion
* Epilepsy
* Sleep-disturbing environment (noise, newborns, etc.)
* Shift work
* Time difference travel from at least 3 zones more than once a month during the study period
* BMI>30
* Drug use in the 3 months prior to inclusion (including caffeine addiction at investigator's discretion)
* Weekly alcohol consumption of more than 21 glasses for a man and 14 for a woman (without exceeding 4 glasses per day and with at least one alcohol-free evening during the week)
* Use of alcohol to sleep
* Pregnant, parturient or breastfeeding women / Subject deprived of liberty by administrative or judicial decision / Persons under guardianship or curatorship or adults protected by law according to articles L1121-5 to L1121-8
* Subjects not affiliated with social security
* Subject with psychological and/or linguistic incapacity to understand and follow the constraints of the study
* Participation in another interventional clinical study where the intervention may have an impact on the objective and primary endpoint during the 4 weeks prior to the start of the study.
* A person who has participated in another research study with an exclusion period still in progress at the time of inclusion.
* Subject who would receive more than 4500 euros in compensation for participation in other biomedical research in the 12 months prior to this study
* Subject cannot be contacted in case of emergency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the URGOnight device on the severity of insomnia | Change from Baseline ISI score at 4 months of treatment
  Assessed by the Insomnia Severity Index (ISI) score

SECONDARY OUTCOMES:
Adherence to therapy | During the 4 months of treatment
  Average frequency of use greater than or equal to 12 sessions per month and the number of training interruptions of more than 7 days less than 2, combined to report adherence to therapy
Acceptability assessed through the motivation of the subject | Visit 3 (Day 100)
  Motivation to do the exercises evaluated by a Visual Analog Scale (VAS)
Ease of use perceived by the user | Visit 3 (Day 100)
  Evaluation by a satisfaction questionnaire: comfort, aesthetics, practicality, ...
Learning to control the neurofeedback task | Up to 4 months of treatment
  Measurement of the amplitude in µV² of SMR activity in baseline and during exercises
Performance during neurofeedback exercises | Up to 4 months of treatment
  Progression of URGOnight neurofeedback training scores calculated by the application
Effect of the URGOnight device on subjective sleep efficiency (WASO) | V0 (Day 0), V2 (Day 65) and V4 (Day 114)
  Wake After Sleep Onset (WASO) determined by sleep diary
Effect of the URGOnight device on subjective sleep efficiency (SOL) | V0 (Day 0), V2 (Day 65) and V4 (Day 114)
  Sleep Onset Latency (SOL) determined by sleep diary
Effect of the URGOnight device on subjective sleep efficiency (TST) | V0 (Day 0), V2 (Day 65) and V4 (Day 114)
  Total Sleep Time (TST) determined by sleep diary
Effect of the URGOnight device on subjective sleep efficiency (SE) | V0 (Day 0), V2 (Day 65) and V4 (Day 114)
  Sleep efficiency (SE) determined by sleep diary
Effect of the URGOnight device on objective sleep efficiency (WASO) | V1 (Day 2) and V5 (Day 116)
  Wake After Sleep Onset (WASO) determined by polysomnography
Effect of the URGOnight device on objective sleep efficiency (SOL) | V1 (Day 2) and V5 (Day 116)
  Sleep Onset Latency (SOL) determined by polysomnography
Effect of the URGOnight device on objective sleep efficiency (TST) | V1 (Day 2) and V5 (Day 116)
  Total Sleep Time (TST) determined by polysomnography
Effect of the URGOnight device on objective sleep efficiency (SE) | V1 (Day 2) and V5 (Day 116)
  Sleep efficiency (SE) determined by polysomnography
Effect of the URGOnight device on objective sleep efficiency (Sleep fragmentation index) | V1 (Day 2) and V5 (Day 116)
  Sleep fragmentation index determined by polysomnography
Increase in sleep satisfaction | Up to 4 months of treatment
  Sleep questionnaire in the application (overall score)
Progression of the sleep hygiene | Up to 4 months of treatment
  Sleep hygiene questionnaire in the application (overall score)
Effect of the URGOnight device on quality of life (Daytime sleepiness) | V0 (Day 0) and V5 (Day 116)
  Epworth Sleepiness Scale (ESS) questionnaire
Effect of the URGOnight device on quality of life (Overall perceived improvement) | Visit 5 (Day 116)
  Patient global Impression of Improvement (PGI-I) questionnaire
Maintaining of sleep improvement | V6 (6-month follow-up visit) and V7 (9-month follow-up visit)
  Insomnia Severity Index (ISI) questionnaire
Effect of the URGOnight device on sleep and wakefulness physiology (resting EEG) | V1 (Day 2) and V5 (Day 116)
  Resting electroencephalographic (EEG) test (10-20 min)
Effect of the URGOnight device on sleep physiology (density of sleep zones) | V1 (Day 2) and V5 (Day 116)
  Density of sleep zones by polysomnography
Effect of the URGOnight device on sleep physiology (amplitude of sleep zones) | V1 (Day 2) and V5 (Day 116)
  Amplitude of sleep zones by polysomnography
Effect of the URGOnight device on sleep physiology (time spent in each sleep stages) | V1 (Day 2) and V5 (Day 116)
  Percentage of time spent in each sleep stage determined by polysomnography
Effect of the URGOnight device on wakefulness physiology (time spent in each sleep stages) | V1 (Day 2) and V5 (Day 116)
  Percentage of time spent in each sleep stage determined by polysomnography
Effect of the device on memory | V1 (Day 2), V2 (Day 65) and V5 (Day 116)
  McNair Self-Questionnaire
Effect of the device on anxiety | V1 (Day 2), V2 (Day 65) and V5 (Day 116)
  State-Trait Anxiety Inventory Y-A Form (STAI-YA)
Device safety | Through study completion (an average of 10 months)
  Collection of Adverse Events
Strategies used to get the exercises done | Up to 4 months of treatment
  Collection of the strategy employed (in the application)
Sub-group analysis of all judging criteria based on chronotype | Visit 1 (Day 2)
  HORNE and OBSERG Circadian Typology Questionnaire
Sub-group analysis of all judging criteria based on level of control over technology | Visit 1 (Day 2)
  KUT (One-Dimensional Target Neutral) Locus of Control Questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Pellegrin University Hospital, Bordeaux
  - Grenoble Alpes University Hospital, Grenoble
  - Lille University Hospital, Lille
  - Hôpital Hôtel-Dieu - APHP, Paris